CLINICAL TRIAL: NCT07063147
Title: Improving the Clinical Management of Stable Chest Pain Based on Imaging: a Registry of Transthorcic Echocardiography
Brief Title: TTE Improves Clinical Management of Stable Chest Pain
Acronym: TICM-SCP
Status: Recruiting | Type: Observational
Sponsor: Tianjin Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhou Jia, Principal Investigator, Tianjin Chest Hospital
Other Study IDs: 2025KY-019-01
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Transthorcic Echocardiography; Stable Angina Pectoris; Coronary Artery Disease; Major Adverse Cardiac Events; Invasive Coronary Angiography
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TTE
  Interventions: Diagnostic Test: TTE

INTERVENTIONS:
Diagnostic Test: TTE — All patients underwent TTE according to established guidelines and local institutional protocols. The imaging data were evaluated using different image post-processing software to comprehensively analyse anatomical, functional and histological information of coronary.

SUMMARY:
The investigator aims to prospectively enroll patients who were referred for transthorcic echocardiography (TTE) for the assessment of stable chest pain (SCP) suspected of obstructive coronary artery disease (CAD). All patients underwent TTE according to established guidelines and local institutional protocols. This study will determine if TTE-based imaging evaluation can provide more informaton to improve clinical management for SCP, including fewer MACE and better decision-making of downstream investigations and therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patients with SCP suspected of obstructive CAD.
* referred for TTE for the assessment of SCP.
* ≥18 years of age.
* signed informed consent.

Exclusion Criteria:

* acute coronary syndromes
* previous CAD or coronary revascularization
* nonsinus rhythm
* cardiomyopathy, valvular disease, congenital heart disease or left cardiac insufficiency because of other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were referred for TTE for the assessment of SCP suspected of CAD.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 10 years

SECONDARY OUTCOMES:
Invasive coronary angiography | 10 years
  Invasive coronary angiography occurred at follow-up after TTE, attributed to TTE results or unplanned.
Medication prescription | 10 years
  Change for medication prescription of antiplatelet agents, anti-ischemic drugs, lipid-lowering agents, angiotensin-converting enzyme inhibition and so on, attributed to TTE results or unplanned,
Coronary revascularization | 10 years
  PTCA, PCI or CABG occurred at follow-up after TTE, attributed to TTE results or unplanned.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Chest Hospital, Tianjin, China